CLINICAL TRIAL: NCT07377539
Title: A Double-Blind, Sponsor-Unblinded, Randomized, Placebo-Controlled Study of the Safety, Tolerability, and Pharmacokinetics of Single-Ascending Doses of JZP047 and an Open-Label Food Effect Study of JZP047 in Healthy Male and Female Participants
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Food Effect of JZP047 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Jazz Pharmaceuticals Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: JZP047-101
Record Dates: First submitted 2026-01-21; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; JZP047

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: JZP047 (Experimental): Healthy participants who are randomized to JZP047.
  Interventions: Drug: JZP047
- Part A: Placebo (Placebo Comparator): Healthy participants who are randomized to placebo.
  Interventions: Other: Placebo
- Part B: JZP047 (Experimental): Healthy participants who will receive JZP047.
  Interventions: Drug: JZP047

INTERVENTIONS:
Drug: JZP047 — Single dose
  Arms: Part A: JZP047; Part B: JZP047
Other: Placebo — Single dose
  Arms: Part A: Placebo

SUMMARY:
This is a Phase 1, double-blind, sponsor-unblinded, randomized, placebo-controlled study designed to characterize the safety, tolerability, and PK of JZP047 in healthy participants following single-ascending doses of study intervention. Additionally, the effect of food on PK following a single dose of JZP047 will be assessed through comparison of PK between the fed and fasted states.

DETAILED DESCRIPTION:
The study will consist of 2 parts: a single-dose ascending part (Part A [SAD] and a single dose under fed conditions part (Part B [Fed PK]).

The study design for Part A will be double-blind, sponsor-unblinded, randomized, and placebo-controlled. Part B, the single dose under fed conditions, will have an open-label study design.

Part A will characterize safety, tolerability, and PK following single doses of JZP047 and matching placebo in healthy male and female participants. Part B will explore the effect of food on a single dose of JZP047 in healthy male and female participants in the fed state.

ELIGIBILITY:
Participants are eligible to be included in the study only if all of the following criteria apply:

1. Healthy participants 18 to 55 years of age, willing and able to comply with study requirements.
2. Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 120 days after the last dose of study intervention:

   * Refrain from donating sperm.
   * Use contraception/barrier as follows:

     * Use a male condom with female partner and use of an additional highly effective contraceptive method with a failure rate of < 1% per year and should also be advised of the benefit of a female partner using a highly effective method of contraception, as a condom may break or leak, when having sexual intercourse with a woman of childbearing potential (WOCBP) who is currently not pregnant.
     * Agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person.
3. Female participants are eligible to participate if:

   * She is a woman of nonchildbearing potential (WONCBP).
   * Pregnancy testing will be performed prior to administration of study intervention to confirm female participants are not pregnant.

Participants are excluded from the study if any of the following criteria apply:

1. History of or presence of clinically significant medical illness or disorder or have a medical issue that may interfere with absorption, distribution, metabolism, or excretion of drugs..
2. History or presence of clinically significant allergy (other than seasonal allergies that do not require treatment during the study) or clinically significant allergy to adhesive bandages, adhesive dressing, ECG patches, or medical tape.
3. History (within 5 past years) or presence of a diagnosis of alcohol abuse, a substance abuse disorder, known drug dependence, or seeking of treatment for an alcohol- or substance abuse-related disorder.
4. Current diagnosis of or receiving treatment for depression; past (within 5 years) clinically significant major depressive episode.
5. History of suicide attempt, current suicidal risk as determined from history, or presence of active suicidal ideation.
6. Presence of any other condition that will cause a risk to participants if they participate in the study as determined by the investigator.
7. Poor peripheral venous access or history of fainting (or passing out) during blood draws.
8. Use or intent to use any prescription medications or nonprescription drugs (including vitamins, recreational drugs, and dietary or herbal supplements) within 14 days or for 5 half-lives, whichever is longer prior to Check-in and throughout the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-02-03 (Estimated); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting Treatment-emergent Adverse Events (Part A) | Baseline up to Day 90
Number of Participants Reporting Treatment-emergent Adverse Events (Part B) | Baseline up to Day 90
Number of Participants Who Discontinued The Study (Part A) | Baseline up to Day 90
Number of Participants Who Discontinued The Study (Part B) | Baseline up to Day 90
Pharmacokinetic Parameter Maximum Concentration (Part A) | Up to 90 days
Pharmacokinetic Parameter Time to Maximum Concentration and Time Before the Start of Absorption (Part A) | Up to 90 days
Pharmacokinetic Parameter Terminal Elimination Half-life (Part A) | Up to 90 days
Pharmacokinetic Parameter Terminal Elimination Rate Constant (Part A) | Up to 90 days
Pharmacokinetic Parameter Volume of Distribution During Terminal Phase (Part A) | Up to 90 days
Pharmacokinetic Parameter Oral Clearance (Part A) | Up to 90 days
Pharmacokinetic Parameter Area Under the Concentration-Time Curve (Part A) | Up to 90 days
  Area under the concentration-time curve from time 0 to 24 (AUC0-24), 0 to last measurable concentration (AUClast), and 0 to infinity (AUC∞) will be assessed.
Pharmacokinetic Parameter Percentage of The Area Under the Concentration-Time Curve From Time Infinity Due to Extrapolation From The Last Quantifiable Concentration to Time Infinity (Part A) | Up to 90 days

SECONDARY OUTCOMES:
Dose Proportionality of JZP047 Cmax (Part A) | Up to 90 days
Dose Proportionality of JZP047 AUC0-last and AUC∞ | Up to 90 days
The Effect of Food On The Single Dose PK of JZP047 Cmax | Up to 90 days
The Effect of Food On The Single Dose PK of JZP047 AUC0-last and AUC∞ | Up to 90 days

IPD SHARING:
Plan to Share IPD: No